CLINICAL TRIAL: NCT03881345
Title: Russian Registry of Treatment of Venous Thromboembolism
Brief Title: Ongoing Registry of Treatment of Venous Thromboembolism
Acronym: RRT VTE
Status: Recruiting | Type: Observational
Sponsor: Medalp Private Surgery Clinic (Other)
Collaborators: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Evgeny Ilyukhin, Principal Investigator, Medalp Private Surgery Clinic
Other Study IDs: A002
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Deep Vein Thrombosis; Thromboses, Venous; Thrombosis Embolism; Postthrombotic Syndrome; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Embolism and Thrombosis; Postthrombotic Syndrome; Pulmonary Embolism | interventions — Anticoagulants; Conversion to Open Surgery; Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Anticoagulants — anticoagulation according to the main diagnosis
Procedure: Open surgery — removal of blood clots with open surgery
Procedure: Thrombolysis — removal of blood clots with thrombolysis
Procedure: Venous stenting — elimination of vein obstruction by stenting

SUMMARY:
Ongoing registration of patients with venous thromboembolism treated by means of antithrombotic therapy, thrombolisys, open surgery, endovenous desobstruction and stenting.

DETAILED DESCRIPTION:
Data of patients with VTE treated in different Russian medical centers are entered in a prospective digital database, and continuously updated.

There is planned to conduct prospective randomized, cohort and observational studies on the site of register

ELIGIBILITY:
Inclusion Criteria:

* case of venous thrombosis of a limb or pulmonary embolus

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing any kind of treatment for venous thromboembolism
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2036-03-01 (Estimated); Study Completion 2036-03-01 (Estimated)

PRIMARY OUTCOMES:
Veins patency | Baseline, 3 and 12 months post-intervention
  Change in patency target veins assessed by duplex ultrasonography in different follow up periods due to different treatment methods

SECONDARY OUTCOMES:
Postthrombotic syndrome | Baseline, 3 and 12 months post-intervention
  the presence and severity of postthrombotic syndrome on the Villalta scale
QoL SF-36 | Baseline, 3 and 12 months post-intervention
  Change in Quality of Life (QoL), assessed by "Short form 36" health survey (SF-36). Total scale range: from 0 to 800. SF-36 consists of 8 subscales. Each subscale range: 0 - 100. Subscales are combined using a special algorithm described in the instructions for the SF-36. For total scale the higher value represent the worse QoL.
QoL AVVQ | Baseline, 3 and 12 months post-intervention
  Change in Quality of Life (QoL), assessed by "Aberdeen Varicose Vein Questionnaire" (AVVQ). The AVVQ is a disease-specific QoL questionnaire aimed at venous disease. Total scale range: from 0 to 100, where the higher score represent worse QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Russian Registry of Treatment of Venous Thromboembolism (RRT VTE) — http://vte.venousregistry.org/index.php
- See also: Russian Phlebological Association (RPA) — https://phlebounion.ru/en